CLINICAL TRIAL: NCT02138214
Title: Thyroid Gland Removal With or Without Central Lymph Node Dissection in Treating Patients With Node Negative Thyroid Cancer
Brief Title: Central Neck Dissection in Patients With Clinical Node Negative Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW13115; NCI-2014-00833 (Registry Identifier: NCI Trial ID); UW13115 (Other: University of Wisconsin Carbone Cancer Center); R01CA176911 (NIH); 2014-0391 (Other: UW-Madison Health Sciences IRB); A539700 (Other: UW Madison); SMPH\SURGERY\SURGERY (Other: UW Madison)
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-02

CONDITIONS: Stage I Papillary Thyroid Cancer; Stage II Papillary Thyroid Cancer; Stage III Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary | interventions — Thyroidectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (no CND) (Experimental): Patients undergo total thyroidectomy alone.
  Interventions: Procedure: Thyroidectomy; Other: Quality-of-life assessment
- Arm II (CND) (Experimental): Patients undergo total thyroidectomy with ipsilateral prophylactic CND.
  Interventions: Procedure: Thyroidectomy; Procedure: entral lymph node dissection (CLND); Other: Quality-of-life assessment
- Arm III (SOC) (Active Comparator): Patients who are not eligible for randomization into Arm I or Arm II, Standard of Care (SOC) group. No specific trial intervention, treated as per patient and physician preference
  Interventions: Other: Quality-of-life assessment

INTERVENTIONS:
Procedure: Thyroidectomy — Undergo total thyroidectomy
  Arms: Arm I (no CND); Arm II (CND)
Procedure: entral lymph node dissection (CLND) — Undergo total thyroidectomy with ipsilateral prophylactic CND
  Arms: Arm II (CND)
Other: Quality-of-life assessment — Voice evaluation, interviews, ancillary studies

SUMMARY:
This phase II trial studies how well thyroid gland removal with or without central lymph node dissection works in treating patients with thyroid cancer or suspected thyroid cancer that has not spread to the lymph nodes (randomized into Arms I and II). Arms I and II are compared to a standard of care (SOC) Arm III to enable comparison of quality of life among various surgical treatments. Currently, the standard treatment for thyroid cancer is total thyroidectomy, or complete removal of the thyroid. The lymph nodes in the central part of the neck may also be surgically removed, called central lymph node dissection. Prophylactic removal of the lymph nodes may increase the risk of life-threatening complications, and may reduce post-surgery quality of life. It may also prevent the cancer from returning and reduce the need for additional surgery. It is not yet known whether recurrence rates and complication levels are lower after thyroid gland removal alone or with central lymph node dissection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of transient and permanent hypocalcemia

SECONDARY OBJECTIVES:

I. To determine the rate of voice and swallowing problems.

II. To determine the degree to which quality of life (QOL) is compromised.

III. To determine the degree to which accurate quality of life measures can be extracted from patient interview narratives using natural language processing techniques.

IV. To determine clinical recurrence rates.

OUTLINE: Patients are randomized to 1 of 2 treatment arms, if ineligible into a SOC arm.

Arm I: Patients undergo total thyroidectomy alone.

Arm II: Patients undergo total thyroidectomy with ipsilateral prophylactic central neck dissection (CND).

Arm III: Patients ineligible to be randomized into Arm I or II, Standard of Care (SOC) comparator receiving same follow up.

After completion of study treatment, patients are followed up at day 1, 2 and 6 weeks, and 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Pre-operative diagnosis or suspicion of papillary thyroid cancer, usually by fine needle aspiration (FNA)
* No pre-operative evidence of cervical lymph node metastases on neck ultrasound (randomization arms only)
* No evidence of distant metastases
* Ability to read and write in English

Exclusion Criteria:

* Largest papillary thyroid carcinoma < 1 cm in size on ultrasound
* Previous thyroid surgery
* Concurrent active malignancy of another type
* Inability to give informed consent or lacks decision making capacity
* T4 tumor
* Pre-existing vocal cord paralysis
* Chronic neurologic condition which affects voice or swallow (for instance, multiple sclerosis or Parkinson disease)
* Baseline laryngeal pathology that would warrant intervention that could affect voice or swallow function
* Becomes pregnant before surgery or at any time while on study

INTRA-OPERATION EXCLUSION CRITERIA (randomization arms only)

* Evidence of nodal involvement identified in the operating room (OR)
* Failure to confirm diagnosis of cancer in participant

Ages: 21 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2014-06-06 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Sippel, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Knigge MA, Robbins D, Thibeault S, Connor N, Sippel R. Secondary analyses of swallowing efficiency and safety outcomes following thyroidectomy versus thyroidectomy plus prophylactic central neck dissection. Thyroid Res. 2025 Sep 16;18(1):45. doi: 10.1186/s13044-025-00264-5. PMID 40954474
- [Derived] Sippel RS, Robbins SE, Poehls JL, Pitt SC, Chen H, Leverson G, Long KL, Schneider DF, Connor NP. A Randomized Controlled Clinical Trial: No Clear Benefit to Prophylactic Central Neck Dissection in Patients With Clinically Node Negative Papillary Thyroid Cancer. Ann Surg. 2020 Sep 1;272(3):496-503. doi: 10.1097/SLA.0000000000004345. PMID 33759836
- [Derived] Kletzien H, Macdonald CL, Orne J, Francis DO, Leverson G, Wendt E, Sippel RS, Connor NP. Comparison Between Patient-Perceived Voice Changes and Quantitative Voice Measures in the First Postoperative Year After Thyroidectomy: A Secondary Analysis of a Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Nov 1;144(11):995-1003. doi: 10.1001/jamaoto.2018.0309. PMID 29710208
- See also: University of Wisconsin Carbone Cancer Center Homepage — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 117 participants consented. 27 participants were excluded from the study before assignment to arms (15 participants withdrew before surgery, 12 participants did not meet intraoperative inclusion criteria). 90 participants were allocated in 3 arms
Groups:
- Arm II (CND): Patients undergo total thyroidectomy with ipsilateral prophylactic CND.
  Thyroidectomy: Undergo total thyroidectomy
  Central lymph node dissection: Undergo total thyroidectomy with ipsilateral prophylactic CND
  Quality-of-life assessment: Voice evaluation, interviews, ancillary studies
Period: Overall Study
Arm/Group | Arm I (no CND) | Arm II (CND) | Arm III (SOC)
Started | 30 | 30 | 30
Analyzed for Baseline Measures | 30 | 29 | 30
Completed | 30 | 26 | 26
Not Completed | 0 | 4 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 4
Not completed — Screen Failure | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (no CND) | Arm II (CND) | Arm III (SOC) | Total
Number analyzed (Participants) | 30 | 29 | 30 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.10 (1.47) | 50.07 (2.38) | 43.17 (2.68) | 46.40 (1.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 27 | 71
  Male | 7 | 8 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 29 | 29 | 28 | 86
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 30 | 28 | 27 | 85
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 30 | 89

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Transient Hypoparathyroidism, as Defined by a Day 1 Serum Parathyroid Hormone (PTH) Level of < 10 pg/ml
Description: Rate of transient hypoparathyroidism will be assessed in terms of percentage of participants with day 1 serum PTH level of < 10 pg/ml.
Time Frame: Post-operative day 1
Population: 1 participant in the Arm II(CND) was a screen failure. Arm III(SOC) data was not collected for this outcome measure as outcome is a comparison of complication rates between TT and CND arms and does not apply to SOC arm participants. The SOC arm was added later as comparison for the qualitative aims only.
Measure: Number; unit: percentage of participants
Arm/Group | Arm II (CND) | Arm I (no CND)
Number analyzed (Participants) | 29 | 30
percentage of participants | 24.1 | 33.3
Statistical Analysis 1: Comparison: Arm II (CND) vs Arm I (no CND); Test type: Other; p = 0.567, Fisher Exact — p-value threshold for statistical significance is 0.05

2. Primary Outcome: Post-operative Serum Calcium (mg/dL) at Day 12
Description: Post-operative serum calcium (mg/dL) at Day 12
Time Frame: At day 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Arm II (CND) | Arm I (no CND)
Number analyzed (Participants) | 29 | 30
mg/dL | 9.39 (0.12) | 9.13 (0.1)
Statistical Analysis 1: Comparison: Arm II (CND) vs Arm I (no CND); Test type: Other; p = 0.110, t-test, 2 sided

3. Primary Outcome: Total Calcium Consumption in First 2 Weeks
Description: Total calcium consumption in first 2 weeks (total mg). Participants were given calcium symptom logs in which to record their calcium consumption between surgery and their first preoperative follow up appointment, approximately two week.
Time Frame: 2 weeks after surgery
Population: 19 participants in CND arm, 22 in 'no CND' arm returned their calcium symptom log to study staff at the end of the postoperative follow-up period. Missing data is due to participants losing/forgetting to return their calcium symptom logs/lack of clarity in their handwritten log entries. This may also have led to limited reliability/accuracy of the data we were able to collect. SOC arm data was not collected as outcome is a comparison of complication rates between TT and CND arms, N/A to SOC arm.
Measure: Mean (Standard Error); unit: mg
Arm/Group | Arm II (CND) | Arm I (no CND)
Number analyzed (Participants) | 19 | 22
mg | 21876.63 (6353.42) | 25470.19 (6592.60)

4. Primary Outcome: Number of Participants With Hypocalcemia Symptoms in First 2 Weeks
Description: Number of participants with hypocalcemia symptoms and symptom severity in first two weeks, as defined by presence of clinically significant symptoms of hypocalcemia.
  Clinically significant symptoms defined as 1 or more episodes of symptoms of hypocalcemia per day for multiple days, symptoms leading to calls to provider for assistance with managing and/or symptoms leading to escalation of dosage of prescribed medications to treat symptoms of hypocalcemia
Time Frame: 2 weeks
Population: In Arm II (CND) 1 participant was lost to screen failure, 1 self-withdrew. Arm III(SOC) data was not collected for this outcome measure as outcome is a comparison of complication rates between TT and CND arms and does not apply to SOC arm participants. The SOC arm was added later as comparison for the qualitative aims only.
Measure: Number; unit: participants
Arm/Group | Arm II (CND) | Arm I (no CND)
Number analyzed (Participants) | 28 | 30
participants | 8 | 6
Statistical Analysis 1: Comparison: Arm II (CND) vs Arm I (no CND); Test type: Other; p = 0.758, Fisher Exact

5. Primary Outcome: Hypocalcemia Symptom Severity Scale (Range of 1-5)
Description: Mean number of occurrences of mild (severity 1 - 2) and severe (severity 3 - 5) hypocalcemia symptoms. Participants were asked to record hypocalcemia symptoms between surgery and first postoperative follow-up at approximately two weeks in their provided calcium symptom logs and rank severity on scale of 1 (mild) to 5 (severe).
Time Frame: 2 weeks post surgery
Population: Missing data is due to participants losing/forgetting to return their calcium symptom logs/lack of clarity in their handwritten log entries. This may also have led to limited reliability/accuracy of the data we were able to collect. SOC arm data was not collected as outcome is a comparison of complication rates between TT and CND arms, not applicable (N/A) to SOC arm.
Measure: Mean (Standard Error); unit: occurrences
Arm/Group | Arm II (CND) | Arm I (no CND)
Number analyzed (Participants) | 13 | 19
occurrences
  mild symptoms (severity 1 - 2) | 3 (1.49) | 2.50 (0.81)
  severe symptoms (severity 3 - 5) | 3.36 (1.59) | 1.42 (0.73)

6. Primary Outcome: Percentage of Participants That Required Calcium and Calcitriol at Month 6
Description: Requirement for calcium and calcitriol at Month 6 (or, if laboratory values at visit reveal calcium < 8 mg/dL and PTH <15 pg/ml)
Time Frame: At Month 6
Population: In Arm II (CND) 1 participant was lost to screen failure, 1 self-withdrew, 1 was lost to follow up. Arm III(SOC) data was not collected for this outcome measure as outcome is a comparison of complication rates between TT and CND arms and does not apply to SOC arm participants. The SOC arm was added later as comparison for the qualitative aims only.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm II (CND) | Arm I (no CND)
Number analyzed (Participants) | 27 | 30
Participants | 0 | 3
Statistical Analysis 1: Comparison: Arm II (CND) vs Arm I (no CND); Test type: Other; p = 0.236, Fisher Exact

7. Primary Outcome: Post-operative Serum PTH (pg/ml) at Month 6
Time Frame: At Month 6
Population: as for outcome 6
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Arm II (CND) | Arm I (no CND)
Number analyzed (Participants) | 27 | 30
pg/mL | 45.62 (4.6) | 44.24 (4.97)
Statistical Analysis 1: Comparison: Arm II (CND) vs Arm I (no CND); Test type: Other; p = 0.759, t-test, 2 sided

8. Primary Outcome: Post-operative Serum Calcium Level at Month 6
Description: Post-operative serum calcium (mg/dL) at Month 6
Time Frame: At Month 6
Population: as for outcome 6
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Arm II (CND) | Arm I (no CND)
Number analyzed (Participants) | 27 | 30
mg/dL | 9.12 (0.08) | 8.98 (0.13)
Statistical Analysis 1: Comparison: Arm II (CND) vs Arm I (no CND); Test type: Other; p = 0.400, t-test, 2 sided

9. Secondary Outcome: Rate of Transient and Permanent Hypocalcemia
Description: The rate of transient and permanent hypocalcemia will be determined by assessing the following:
  I. Post-operative serum calcium (mg/dl) and PTH (pg/ml) at Day 12 and Month 6 II. Total calcium consumption in first 2 weeks (total gm) III. Hypocalcemia symptoms in first 2 weeks (average episodes/day) IV. Hypocalcemia symptom severity scale (range 1-5) V. Requirement for calcium and calcitriol at Month 6 (or, if laboratory values at visit reveal calcium < 8 mg/dL and PTH < 15 pg/ml
  Data will be analyzed using the methods described above.
Time Frame: Post-operative day 1 - Month 6
Reporting Status: Not Posted

10. Secondary Outcome: Rate of Voice and Swallowing Problems
Description: The rate of voice and swallowing problems will be determined by assessing the following:
  I. Phonation threshold pressure, in centimeters of water II. Dysphonia severity index (DSI) score (+5 to -5) III. Grade Roughness Breathiness Asthenia Strain (GRBAS) score (0-3) IV. Voice quality parameters as measured by Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) (0-100 on visual analog scale) V. Vocal fold vibratory and movement parameters as measured by stroboscopy assessment (1-4) VI. Glottal function index score VII. Penetration-Aspiration score as measured by videofluoroscopic swallow study (0-8)
  Data will be analyzed using the methods described above.
Time Frame: Post operative day 1 - up to 1 year
Reporting Status: Not Posted

11. Secondary Outcome: Degree to Which Quality of Life (QOL) is Compromised
Description: The degree to which quality (QOL) is compromised will be determined by assessing the following:
  I. Short Form Health Survey (SF-12) Mental Composite Scale (MCS) score II. Short Form Health Survey (SF-12) Physical Composite Scale (PCS) score III. European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Core-30 (C30) score IV. Thyroid Cancer Specific Quality of Life (ThyCA-QOL) score V. 10-item Eating Assessment Tool (EAT-10) dysphagia inventory score VI. Voice Handicap Index (VHI) score VII. Themes and codes from interview transcripts assessed using qualitative research methods
  Data will be analyzed using the methods described above.
Time Frame: Post-operative day 1 - up to 1 year
Reporting Status: Not Posted

12. Secondary Outcome: Clinical Recurrence Rates
Description: Clinical recurrence rates will be determined by assessing the following:
  I. Percent of patients with a recombinant thyroid-stimulating hormone (rTSH) stimulated thyroglobulin level < 1 ng/ml one year after surgery II. Unstimulated thyroglobulin level prior to beginning week 6 radioactive iodine treatment III. Stimulated thyroglobulin at the time of week 6 radioactive iodine treatment IV. Incidence of unstimulated thyroglobulin > 1 ng/mL at 6 months V. Incidence of stimulated thyroglobulin > 2 ng/mL at 1 year VI. Incidence of biopsy-proven disease identification on neck ultrasound or iodine-131 (I-131) uptake up to 5 years post-surgery
  Data will be analyzed using the methods described above.
Time Frame: Week 6 - up to 5 years
Reporting Status: Not Posted

13. Secondary Outcome: Degree to Which Accurate Quality of Life (QOL) Measures Can be Extracted From Patient Interview Narratives Using Natural Language Processing Techniques
Description: The degree to which accurate quality of life (QOL) measures can be extracted from patient interview narratives using natural language process techniques will allow for the development of computer algorithms that convert patient narrative text into simple quality of life measures. Data will be analyzed using the methods described above.
Time Frame: Post-operative day 1 - up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm I (no CND) | Arm II (CND) | Arm III (SOC)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 23/30 | 25/29 | 9/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (no CND) (N=30) | Arm II (CND) (N=29) | Arm III (SOC) (N=30)
biochemical hypopcalcemia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) — Serum calcium <8.0 mg/dL at any single time point
symptomatic hypoparathyroidism (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 1 (1) — * The need for calcium or calcitriol to prevent symptoms of hypocalcemia * Evidenced by paresthesias and/or muscle cramps which are improved or relieved with calcium * Requiring frequent treatment with calcium and vitamin D
nerve injury (Injury, poisoning and procedural complications) | 12 (12) | 7 (7) | 3 (3) — Injury to or dysfunction of the recurrent laryngeal nerve (RLN) or superior laryngeal nerve (SLN) as complication of thyroid surgery
significant voice changes not otherwise characterized (Injury, poisoning and procedural complications) | 11 (11) | 7 (7) | 2 (2) — If patient needs further voice evaluations beyond two-week time point, this is indication of significant voice change(s)
biochemical hypoparathyroidism (Injury, poisoning and procedural complications) | 9 (9) | 8 (8) | 3 (3) — Serum PTH level <10 pg/ml
symptomatic hypocalcemia (Injury, poisoning and procedural complications) | 4 (4) | 6 (6) | 2 (2) — Significant symptomatic hypocalcemia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT02138214/Prot_SAP_000.pdf